CLINICAL TRIAL: NCT05451069
Title: Combined Neurofilament Light Chain ,Chitinase-3 Like-1 Protein Levels and Tolerogenic Plasmacytoid Dendritic Cells in Defining Disease Course in Multiple Sclerosis Patients
Brief Title: Neurofilament Light Chain ,Chitinase-3 Like-1 Proteins and Plasmacytoid Dendritic Cells in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bassant Rashad, Principal Investigator (Assistant Lecturer of Clinical pathology), Assiut University
Other Study IDs: Multiple Sclerosis markers
Record Dates: First submitted 2022-06-26; First posted 2022-07-11 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood samples(EDTA and Serum) Cerebrospinal fluid(CSF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple sclerosis patients: MS patients according to 2017 Macdonald criteria
  Interventions: Diagnostic Test: Neurofilament Light Chain ,Chitinase-3 Like-1 Protein Levels and Tolerogenic plasmacytoid Dendritic Cells
- Non Multiple sclerosis persons: Control persons
  Interventions: Diagnostic Test: Neurofilament Light Chain ,Chitinase-3 Like-1 Protein Levels and Tolerogenic plasmacytoid Dendritic Cells

INTERVENTIONS:
Diagnostic Test: Neurofilament Light Chain ,Chitinase-3 Like-1 Protein Levels and Tolerogenic plasmacytoid Dendritic Cells — 1. Serum and CSF levels assay of NfL and CHI3L1 using the enzyme linked immunosorbent assay kits (ELISA).
  2. Peripheral blood mononuclear cells (PBMC) will be obtained by Ficoll-Hypaque gradient. plasmacytoid dendritic cells will be identified in (CSF) and (PBMN) based on their selective expression of surface antigen (cluster of differentiation 303) CD303, named blood dendritic cells antigen 2 (BDCA-2).Antihuman antibodies: BDCA-2, HLA-DR , CD274 , HLA-G and CCR7 for identification of tolerogenic plasmacytoid dendritic cells using flowcytometry.

SUMMARY:
Multiple sclerosis (MS) is an autoimmune neurodegenerative disease characterized by demyelination and neurodegeneration of the central nervous system (CNS) . Current diagnostic criteria and management depend on MRI, clinical status, and oligoclonal immunoglobulin g bands . These markers often fail to predict relapse, progression and therapy response .There is an increased need to identify biomarkers for clinical endpoints .

One of the hallmark features of MS is axonal damage which associated with brain and cervical atrophy.Nf levels indicate the extent of axonal damage. Neurofilaments are composed of four subunits: neurofilament light polypeptides (NfL) is the most abundant and soluble and it is highly sensitive to neurodegenerative processes .

Chitinase 3-like 1 (CHI3L1) is expressed in astrocytes in the brain tissue of MS patients . CHI3L1 plays a role as prognostic biomarker in patients with MS. CHI3L1 cerebrospinal fluid levels were associated correlated with disease activity and neurological disability.

Dendritic cells (DCs) are highly specialized antigen-presenting cells with a key role in activating and preventing CNS immune-mediated damage in MS . Dendritic cells express Human Leukocyte Antigen-antigen D Related (HLA-DR) . Plasmacytoid dendritic cells characterized by the expression of blood dendritic cells antigen-2 (BDCA-2) .Plasmacytoid dendritic cells are present in the cerebrospinal fluid (CSF), leptomeninges and demyelinating lesions of patients with MS . Plasmacytoid dendritic cells also exhibit up-regulation of chemokine (CCR7C) expression. It was demonstrated increased amounts of chemokine CCR7 in the CSF from MS patients during relapses .CCR7 controls migration and functional activity of regulatory T cells and plays an important role in the establishment of tolerance .

Tolerogenic DCs (TolDCs) present an intermediate phenotype between immature dendritic cells (iDCs) and mature dendritic cells (mDCs) regarding costimulatory molecules, a pronounced shift toward anti-inflammatory . TolDCs exhibit tolerogenic molecules such as HLA-G and CD274 [programmed death-ligand 1 (PD-L1)] either in peripheral blood or in CSF. These characteristics lead to T cell clonal anergy and T cell unresponsiveness due to Ag presentation in the presence of low co-stimulation .We aim to investigate the role of NfL,(CHI3L1) and markers of plasmacytoid dendritic cells in MS.

ELIGIBILITY:
Inclusion Criteria: 1-MS patients diagnosis 2017 McDonald criteria. 2-Patients age 20-60 years 3-All males and female patients. 3-Willingness and ability to comply with the protocol. 4-Written informed consent given by the patient before the beginning of any study-related procedure, 5-Non-MS control matched age and sex persons

Exclusion Criteria:1-patients with Intracranial space-occupying lesion. 2-Abnormal intracranial pressure due to increased CSF pressure or Arnold-Chiari malformation.

3-Anticoagulant medication, coagulopathies and uncorrected bleeding diathesis. 4-Congenital spine abnormalities. 5-Local skin infection at the puncture site. 6-Not fulfill Macdonald criteria.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 21 MS patients and 21 non-MS control perons.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-07-25 (Estimated); Study Completion 2025-07-27 (Estimated)

PRIMARY OUTCOMES:
Levels of different markers in MS diagnosis | 2 years
  The changes of levels of NfL and CHI3L1 using ELISA kits and its correlation with the expression of identification markers of plasmacytoid dendritic cells and its activity (HLA-DR, BDCA-2, ,CCR7C ,HLA-G and CD274) using flowcytometry in different clinical presentations of MS in consistent with MRI findings.

SECONDARY OUTCOMES:
Different samples levels in MS diagnosis | 2 years
  Changes of levels of NfL and CHI3L1 using ELISA kits and markers of plasmacytoid dendritic using flowcytometry between blood and CSF samples of MS diagnosis.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reich DS, Lucchinetti CF, Calabresi PA. Multiple Sclerosis. N Engl J Med. 2018 Jan 11;378(2):169-180. doi: 10.1056/NEJMra1401483. No abstract available. PMID 29320652
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Hakansson I, Tisell A, Cassel P, Blennow K, Zetterberg H, Lundberg P, Dahle C, Vrethem M, Ernerudh J. Neurofilament light chain in cerebrospinal fluid and prediction of disease activity in clinically isolated syndrome and relapsing-remitting multiple sclerosis. Eur J Neurol. 2017 May;24(5):703-712. doi: 10.1111/ene.13274. Epub 2017 Mar 6. PMID 28261960
- [Background] Ehrenberg AJ, Khatun A, Coomans E, Betts MJ, Capraro F, Thijssen EH, Senkevich K, Bharucha T, Jafarpour M, Young PNE, Jagust W, Carter SF, Lashley T, Grinberg LT, Pereira JB, Mattsson-Carlgren N, Ashton NJ, Hanrieder J, Zetterberg H, Scholl M, Paterson RW. Relevance of biomarkers across different neurodegenerative diseases. Alzheimers Res Ther. 2020 May 13;12(1):56. doi: 10.1186/s13195-020-00601-w. PMID 32404143
- [Background] Ferreira-Atuesta C, Reyes S, Giovanonni G, Gnanapavan S. The Evolution of Neurofilament Light Chain in Multiple Sclerosis. Front Neurosci. 2021 Apr 6;15:642384. doi: 10.3389/fnins.2021.642384. eCollection 2021. PMID 33889068
- [Background] Ziemssen T, Akgun K, Bruck W. Molecular biomarkers in multiple sclerosis. J Neuroinflammation. 2019 Dec 23;16(1):272. doi: 10.1186/s12974-019-1674-2. PMID 31870389
- [Background] Gisslen M, Price RW, Andreasson U, Norgren N, Nilsson S, Hagberg L, Fuchs D, Spudich S, Blennow K, Zetterberg H. Plasma Concentration of the Neurofilament Light Protein (NFL) is a Biomarker of CNS Injury in HIV Infection: A Cross-Sectional Study. EBioMedicine. 2015 Nov 22;3:135-140. doi: 10.1016/j.ebiom.2015.11.036. eCollection 2016 Jan. PMID 26870824
- [Background] Disanto G, Barro C, Benkert P, Naegelin Y, Schadelin S, Giardiello A, Zecca C, Blennow K, Zetterberg H, Leppert D, Kappos L, Gobbi C, Kuhle J; Swiss Multiple Sclerosis Cohort Study Group. Serum Neurofilament light: A biomarker of neuronal damage in multiple sclerosis. Ann Neurol. 2017 Jun;81(6):857-870. doi: 10.1002/ana.24954. PMID 28512753
- [Background] Kusnierova P, Zeman D, Hradilek P, Zapletalova O, Stejskal D. Determination of chitinase 3-like 1 in cerebrospinal fluid in multiple sclerosis and other neurological diseases. PLoS One. 2020 May 21;15(5):e0233519. doi: 10.1371/journal.pone.0233519. eCollection 2020. PMID 32437412
- [Background] Comabella M, Deutschmann C, Midaglia L, Schierack P, Martinez J, Roggenbuck D, Montalban X. Chitinase 3-like 1 is not a target antigen in patients with multiple sclerosis. Mult Scler. 2021 Aug;27(9):1455-1457. doi: 10.1177/1352458520980141. Epub 2020 Dec 17. PMID 33327838
- [Background] Piacente F, Bottero M, Benzi A, Vigo T, Uccelli A, Bruzzone S, Ferrara G. Neuroprotective Potential of Dendritic Cells and Sirtuins in Multiple Sclerosis. Int J Mol Sci. 2022 Apr 14;23(8):4352. doi: 10.3390/ijms23084352. PMID 35457169
- [Background] Florez-Grau G, Zubizarreta I, Cabezon R, Villoslada P, Benitez-Ribas D. Tolerogenic Dendritic Cells as a Promising Antigen-Specific Therapy in the Treatment of Multiple Sclerosis and Neuromyelitis Optica From Preclinical to Clinical Trials. Front Immunol. 2018 May 31;9:1169. doi: 10.3389/fimmu.2018.01169. eCollection 2018. PMID 29904379
- [Background] Passeri L, Marta F, Bassi V, Gregori S. Tolerogenic Dendritic Cell-Based Approaches in Autoimmunity. Int J Mol Sci. 2021 Aug 5;22(16):8415. doi: 10.3390/ijms22168415. PMID 34445143
- [Background] Longhini AL, von Glehn F, Brandao CO, de Paula RF, Pradella F, Moraes AS, Farias AS, Oliveira EC, Quispe-Cabanillas JG, Abreu CH, Damasceno A, Damasceno BP, Balashov KE, Santos LM. Plasmacytoid dendritic cells are increased in cerebrospinal fluid of untreated patients during multiple sclerosis relapse. J Neuroinflammation. 2011 Jan 7;8(1):2. doi: 10.1186/1742-2094-8-2. PMID 21214939